CLINICAL TRIAL: NCT06820333
Title: The Clinical Impact and Prognostic Value of [18F] PSMA-1007 Imaging for Primary Staging of Prostate Cancer: Real-world Evidence From a Monocentric, Prospective Observational Study
Brief Title: Impact of [18F] PSMA-1007 Imaging for Primary Staging of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Emil Novruzov, Dr. med., Heinrich-Heine University, Duesseldorf
Other Study IDs: 2024-3103
Record Dates: First submitted 2025-01-16; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PSMA; PSMA-PET; PSMA PET/CT; Primary Staging
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The introduction of PSMA diagnostics and therapy has fundamentally changed the treatment management of prostate cancer and has significantly replaced other clinical and radiological diagnostic methods. As a result, 18F-PSMA-1007 (Radelumin®) was approved in Germany and several EU countries, most recently in Germany in 01/2024, for use in primary staging of high-risk prostate cancer and re-staging in the context of biochemical recurrence (BCR). This could be seen as a milestone in the management of prostate cancer and will significantly promote the widespread use of PSMA-PET diagnostics in the coming years.

The investigators now intend to prospectively generate evidence-based data in everyday clinical practice with this so-called Real-World-Evidence (RWE) study. The planned study will enable us to analyze the diagnostic accuracy of Radelumin® in more detail under everyday conditions, whereby dedicated examinations of certain subgroups and the prospective generation of a complete, high-quality database for the future use of artificial intelligence (AI) will be made possible.

DETAILED DESCRIPTION:
Depending on the study design and definition of the patient population, the detection rate of pelvic lymph nodes in particular using PSMA imaging is reported to be >80%. The results of the studies thus demonstrate a superior diagnostic accuracy compared to previous methods as well as a significant influence of PSMA imaging on the clinical course. Radelumin® was approved on the basis of these promising results from numerous retrospective studies and the prospective, randomized approval study.

Nevertheless, it should be noted that the results derived from such data generally deviate from the data in everyday clinical practice for various reasons. Furthermore, the retrospectively planned studies show multiple general weaknesses, whereby the prospective randomized approval studies also show a priori weaknesses. These result from a very limited observation phase and the lack of long-term data, despite good planning with a high power, a small number of patients and the targeted homogeneity of the patient population. In the context of a real-world evidence study, which focuses on routine clinical care, the above-mentioned disadvantages are compensated for by long-term observation, a considerably larger patient population and a realistic patient mix.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Planned [18F]PSMA-1007 PET/CT examination in patients with a first diagnosis of prostate cancer
* Informed consent

Exclusion Criteria:

- Examinations with limited assessability due to technical errors, such as imaging artifacts.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biologically male patients are valid study participants because of the disease
Study Population: biologically male patients with biopsy-proven or highly suspected prostate cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy and Prognostic Value of [18F]PSMA-1007 PET/CT in Primary Staging of Prostate Cancer | Interim analyses will be performed annually, with a final analysis at 5 years.
  1. The primary outcome will assess the diagnostic accuracy of [18F]PSMA-1007 PET/CT by comparing its sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) against histopathological confirmation or composite clinical follow-up as the reference standard.
  2. The prognostic value will be evaluated by analyzing the association between baseline PSMA PET/CT-derived parameters (e.g., SUVmax, tumor burden, lesion distribution) and oncological outcomes, including biochemical recurrence-free survival and progression-free survival.
  3. Quantitative PET parameters will be extracted using a standardized semi-automated segmentation method, and survival analysis will be conducted using Kaplan-Meier estimates and Cox proportional hazards models.

SECONDARY OUTCOMES:
Correlation of PET Parameters with Clinical and Pathological Features Description | Evaluated at 1-year, 2-year, and 5-year follow-up.
  1. The correlation between PET-derived quantitative parameters (SUVmax, metabolic tumor volume [MTV], total lesion PSMA expression [TLPE]) and clinical/pathological factors (Gleason Score, PSA level, tumor stage, lymph node involvement) will be assessed.
  2. The proportion of patients whose management plan (e.g., radical prostatectomy, radiotherapy, systemic therapy) changed due to PSMA PET/CT findings compared to conventional imaging. Measured by documenting pre- and post-imaging treatment plans and analyzing changes in therapeutic strategies.
  3. The relationship between baseline PSMA PET/CT findings and biochemical recurrence free survival (BRFS) will be analyzed using Kaplan-Meier survival analysis and Cox proportional hazards modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Lars Giesel, Prof. Dr., Medical Doctor, Study Chair — Department of Nuclear Medicine, Medical Faculty and University Hospital Duesseldorf, Heinrich-Heine-University Duesseldorf
Locations (1):
- Heinrich Heine University, Medical Faculty, University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
At a reasoble request, the study data would be provided.